CLINICAL TRIAL: NCT04835961
Title: This Study Will Record the Use of Budesonide / Formoterol Either as Maintenance Treatment or / or as Needed According to Standard Clinical Practice and at the Discretion of the Treating Physician.
Brief Title: AdditioN of Fixed Dose Combination (FDC) Of Budesonide/Formoterol Via Elpenhaler® Device in Greek Patients With asThma accΟrding to Standard Clinical Practice.
Acronym: NOTOS
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-BUDFOR-EL-127
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: asthma; as needed treatment; maintenance treatment
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Maintenace and As needed — This study will record the use of budesonide / formoterol either as maintenance treatment or / or as needed according to standard clinical practice and at the discretion of the treating physician.

SUMMARY:
The budesonide / formoterol combination can be used both as a maintenance treatment and as a maintenance and relief therapy (MART) where in the latter there is also anti-inflammatory action in contrast to the use of SABA. This anti-inflammatory and soothing effect has been recognized by the Global Initiatives for Asthma (GINA) guidelines and is recommended as a palliative treatment for all types of asthma severity versus Short Acting Beta Agonists (SABA).

Test results have shown that the invoked budesonide / formoterol combination therapy had a similar (not lower) effect on the annual exacerbation rate, with lower exposure to ICS compared to regular maintenance therapy with inhaled corticosteroids (ICS), although budesonide / formoterol therapy appeared to was inferior to ongoing asthma control. Another study showed no inferiority of the stable budesonide / formoterol combination compared to maintenance ICS plus the required SABA dosing regimen in reducing the annual severe exacerbation rate in patients with mild asthma.

Patients receiving budesonide / formoterol as adjunctive therapy or as maintenance therapy experienced a reduced incidence of exacerbations including asthma-related SAEs, compared with patients receiving long acting beta agonists (LABAs) or SABAs as sedatives, ICS or ICS / LA terbutaline or salbutamol. Studies have shown that patients spent more days without palliative care, indicating a significant reduction in reliance on palliative care while improving both disease control and daily functioning and well-being. Asthma symptoms and nocturnal awakening were significantly reduced, and FEV1 levels before and after treatment showed significant improvement in lung function and quality of life as shown by the AQLQ-S questionnaire score. In addition, ICS / LABA therapy as a palliative or maintenance treatment appears to be well tolerated and reduces the risk of severe exacerbations following exposure to high doses of SABA which may mask the worsening of inflammation.

The meta-analysis of Rogliani et. al. showed that low dose (LD) to medium dose (MD) ICS / LABA MART was as effective as HD ICS / LABA and SABA as needed treatments in reducing the risk of severe asthma exacerbations and that MART was generally more effective than low dose LD ICS / LABA + as needed LABA or SABA, or ICS / LABA as needed or ICS + as needed SABA treatments. The efficacy of ICS / LABA as needed treatment in the risk of severe exacerbation was significantly higher than ICS + as needed SABA treatment but not ICS / LABA + as needed SABA in patients with mild to severe asthma. LD to MD MART and HD ICS / LABA + as needed SABA were equally effective (P> 0.05) in improving PEF, and more effective (P <0.05) than LD ICS / LABA + as needed SABA or LABA, ICS / LABA as needed, ICS + SABA as needed, and SABA as needed. Administration of ICS / LABA as purely invasive use significantly improved (P <0.05) PEF compared to ICS + SABA as needed, LD ICS / LABA + SABA as needed, and SABA as needed treatments. MART improved lung function and disease control compared to other invasive therapies in patients with moderate asthma. In contrast, in patients with moderate to severe asthma, LD to MD MART was partially more effective than other invasive therapies in improving lung function and controlling asthma. No differences were found in the safety profile which was measured as the risk of occurrence of YOU.

The combination of budesonide / formoterol as maintenance therapy and as-needed palliative care could improve overall asthma control without the need for additional palliative care.

DETAILED DESCRIPTION:
Pulmoton® is an inhaled combination of budesonide and formoterol fumarate dihydrate in doses of 100 / 6mcg, 200 / 6mcg, 400/12 mcg, administered by Elpenhaler®, a powder inhaler developed in doses developed by the ELPEN. It has been approved as a bronchodilator in the treatment of asthma where combination therapy (ICS / LABA) is appropriate in patients who are not adequately controlled with inhaled corticosteroids and rely on short-acting inhaled β2-stimulants or in patients already satisfactorily controlled with both corticosteroids. long-acting β2-stimulants.

Pulmoton® is not recommended for the initial treatment of asthma. The dosage of the individual components of Pulmoton® is separate and must be adjusted according to the severity of the condition. This should be taken into account, not only when starting treatment with stable combination products, but also when adjusting the maintenance dosage.

The dose should be adjusted to the lowest possible, by which effective control of symptoms is achieved and maintained. Patients should be re-evaluated regularly by their physician so that the dose of Pulmoton® they receive remains the best possible. When long-term control of symptoms is achieved with the lowest recommended dose, then in the next step only the inhaled corticosteroid can be tested.

There are two alternatives to treating asthma with Pulmoton®:

A. Pulmoton® Maintenance Therapy: Pulmoton® is taken as a regular maintenance treatment along with a separate rapid-acting bronchodilator to relieve symptoms.

B. Pulmoton® Maintenance and Relief Therapy: Pulmoton® is also taken as regular maintenance and invocative treatment for symptoms.

Further information on the efficacy and safety of the drug under study can be found in the Product Characteristics Summary (SmPC).

Aims of the study The GINA 2020 guidelines recommend, among other things, the symptom-driven use of ICS / LABA (as needed).

This study will record the use of budesonide / formoterol either as maintenance treatment or / or as needed according to standard clinical practice and at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients Newly diagnosed patients with asthma without prior treatment or receiving previous low dose (LD) ICS / LABA treatment, as needed.
* Patients who are not adequately controlled with LD ICS as maintenance therapy and need to have LABA added:

  * or as a maintenance treatment
  * either as maintenance therapy and as an invocation to treat the symptoms.
* Patients who are not adequately controlled with LD or moderate (MD) ICS and LABA doses and need to have ICS / LABA added as an adjunctive therapy to treat the symptoms.
* Consent and compliance with the therapies and study procedures.

Exclusion Criteria:

Patients <18

* Patients with COPD
* Patients with ACO

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients proflle is based on GINA 2020 guidelines that recommend, among other things, the symptom-driven use of inhaled corticosteroids / long-acting β2-stimulants (ICS / LABA) (as needed).
  This study will record the use of budesonide / formoterol either as maintenance treatment or / or as needed according to standard clinical practice and at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 1037 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Asthma control | 6 months
  Asthma control at 3 and 6 months of treatment.

SECONDARY OUTCOMES:
FEV1 | 6 months
  The evaluation of pulmonary function at 3 and 6 months of treatment.
MiniAQLQ questionnaire | 6 months
  The evaluation of Quality of Life at 3 and 6 months of treatment.
FSI-10 questionnaire | 6 months
  Assessing patient satisfaction with the use of the inhalation device

CONTACTS AND LOCATIONS:
Locations (1):
- Sotiria Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Husseini ZW, Gosens R, Dekker F, Koppelman GH. The genetics of asthma and the promise of genomics-guided drug target discovery. Lancet Respir Med. 2020 Oct;8(10):1045-1056. doi: 10.1016/S2213-2600(20)30363-5. Epub 2020 Sep 7. PMID 32910899
- [Result] 1. Global Initiative for Asthma. Gglobal Strategy for Asthma Management and Prevention. (2020) Available from: www.ginasthma.org
- [Result] Jenkins CR, Bateman ED, Sears MR, O'Byrne PM. What have we learnt about asthma control from trials of budesonide/formoterol as maintenance and reliever? Respirology. 2020 Aug;25(8):804-815. doi: 10.1111/resp.13804. Epub 2020 Mar 31. PMID 32237004
- [Result] Lougheed MD, Lemiere C, Ducharme FM, Licskai C, Dell SD, Rowe BH, Fitzgerald M, Leigh R, Watson W, Boulet LP; Canadian Thoracic Society Asthma Clinical Assembly. Canadian Thoracic Society 2012 guideline update: diagnosis and management of asthma in preschoolers, children and adults. Can Respir J. 2012 Mar-Apr;19(2):127-64. doi: 10.1155/2012/635624. PMID 22536582
- [Result] Kaplan AG, Balter MS, Bell AD, Kim H, McIvor RA. Diagnosis of asthma in adults. CMAJ. 2009 Nov 10;181(10):E210-20. doi: 10.1503/cmaj.080006. Epub 2009 Sep 21. No abstract available. PMID 19770241
- [Result] Lemanske RF Jr, Busse WW. Asthma: clinical expression and molecular mechanisms. J Allergy Clin Immunol. 2010 Feb;125(2 Suppl 2):S95-102. doi: 10.1016/j.jaci.2009.10.047. PMID 20176271
- [Result] Bai TR, Vonk JM, Postma DS, Boezen HM. Severe exacerbations predict excess lung function decline in asthma. Eur Respir J. 2007 Sep;30(3):452-6. doi: 10.1183/09031936.00165106. Epub 2007 May 30. PMID 17537763
- [Result] 8. P. Moraitaki, D. Papamichail, N. Georgatotu (2010) Severe Asthma: Definitions, risk factors and phenotype characterization. Pneumon, 23(3):276-292.
- [Result] 9. P. Latsi, M. Gaga (1999) Leukotriene antagonists, a new class of anti-asthmatic drugs. Pneumon, 12 (2): 123-132
- [Result] Muneswarao J, Hassali MA, Ibrahim B, Saini B, Ali IAH, Verma AK. It is time to change the way we manage mild asthma: an update in GINA 2019. Respir Res. 2019 Aug 14;20(1):183. doi: 10.1186/s12931-019-1159-y. PMID 31412856
- [Result] Bateman ED, Reddel HK, O'Byrne PM, Barnes PJ, Zhong N, Keen C, Jorup C, Lamarca R, Siwek-Posluszna A, FitzGerald JM. As-Needed Budesonide-Formoterol versus Maintenance Budesonide in Mild Asthma. N Engl J Med. 2018 May 17;378(20):1877-1887. doi: 10.1056/NEJMoa1715275. PMID 29768147
- [Result] O'Byrne PM, FitzGerald JM, Bateman ED, Barnes PJ, Zhong N, Keen C, Jorup C, Lamarca R, Ivanov S, Reddel HK. Inhaled Combined Budesonide-Formoterol as Needed in Mild Asthma. N Engl J Med. 2018 May 17;378(20):1865-1876. doi: 10.1056/NEJMoa1715274. PMID 29768149
- [Result] Rogliani P, Ritondo BL, Ora J, Cazzola M, Calzetta L. SMART and as-needed therapies in mild-to-severe asthma: a network meta-analysis. Eur Respir J. 2020 Sep 10;56(3):2000625. doi: 10.1183/13993003.00625-2020. Print 2020 Sep. PMID 32430423
- [Result] Buhl R, Kuna P, Peters MJ, Andersson TL, Naya IP, Peterson S, Rabe KF. The effect of budesonide/formoterol maintenance and reliever therapy on the risk of severe asthma exacerbations following episodes of high reliever use: an exploratory analysis of two randomised, controlled studies with comparisons to standard therapy. Respir Res. 2012 Jul 20;13(1):59. doi: 10.1186/1465-9921-13-59. PMID 22816878
- [Result] Zhong N, Lin J, Mehta P, Ngamjanyaporn P, Wu TC, Yunus F. Real-life effectiveness of budesonide/formoterol maintenance and reliever therapy in asthma patients across Asia: SMARTASIA study. BMC Pulm Med. 2013 Apr 4;13:22. doi: 10.1186/1471-2466-13-22. PMID 23557023
- [Result] Lin J, Zhou X, Wang C, Liu C, Cai S, Huang M. Symbicort(R) Maintenance and Reliever Therapy (SMART) and the evolution of asthma management within the GINA guidelines. Expert Rev Respir Med. 2018 Mar;12(3):191-202. doi: 10.1080/17476348.2018.1429921. Epub 2018 Feb 5. PMID 29400090
- [Result] International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use.. ICH harmonized tripartite guideline: Guideline for Good Clinical Practice. J Postgrad Med. 2001 Jan-Mar;47(1):45-50. No abstract available. PMID 11590294
- [Result] 19. World Medical Association Declaration of Helsinki. Ethical principles for Medical Research Involving Human Subjects, Helsinki 1964, amended in Tokyo 1975, Venice 1983, Hong Kong 1989, Somerset West 1996, Edinburgh 2000, Washington DC 2002, Tokyo 2004, Seoul 2008 and Fortaleza 2013.
- [Result] Epstein M; International Society of Pharmacoepidemiology. Guidelines for good pharmacoepidemiology practices (GPP). Pharmacoepidemiol Drug Saf. 2005 Aug;14(8):589-95. doi: 10.1002/pds.1082. No abstract available. PMID 15918159
- [Result] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Result] Grammatopoulou E, Skordilis E, Koutsouki D, Baltopoulos G. An 18-item standardized Asthma Quality of Life Questionnaire-AQLQ(S). Qual Life Res. 2008 Mar;17(2):323-32. doi: 10.1007/s11136-007-9297-y. Epub 2007 Dec 14. PMID 18080214
- [Result] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Result] 25. Grekas N., Athanassiou A., Iskos C., Panagiotakos D., Papataxiarchou A., Porichi O. (2011). Reliability of the FSI-10 questionnaire for the assessment of the usability of drug inhalers in Greek patients. Archives of Hellenic Medicine, 28(2):257-260
- [Result] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666